CLINICAL TRIAL: NCT03129516
Title: Reliability and Validity of the Turkish Version of the Movement Imagery Questionnaire-3
Brief Title: Turkish Version of the Movement Imagery Questionnaire-3
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Burcu Dilek, PT, MS, PhD, Assist Prof, Hacettepe University
Other Study IDs: GO 14/569
Record Dates: First submitted 2017-04-16; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Image, Body
Keywords: imaginary; Turkish version; motor imagery; reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Determining Imaginary levels — Determining the motor imaginary: internal visual, external visual and kinesthetic imagery

SUMMARY:
Motor imagery is the mental representation of movement without any body movement. According to recent studies motor imagery contains three strategies to mentally simulate the movements: internal visual, external visual and kinesthetic imagery. Motor imagery is associated with cortical reorganization and functional improvements and it does not only related with motor performance, it also influces cognitions. Movement Imagery Questionnaire-3 (MIQ-3) is the recent, modified version of the Movement Imagery Questionnaire-Revised, Second Edition and measures imagery ability in terms of ease of imagery.

The aim of this study is to translate MIQ-3 into Turkish and evaluate its test-retest reliability for Turkish-speaking population.

ELIGIBILITY:
Inclusion Criteria:

* age above 18, consenting, with no limitation in mobility or movement disorder

Exclusion Criteria:

* refuse to attend to the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cronbach's Alpha coefficient | 2 years
  Cronbach's Alpha coefficient was used to determine internal consistency of the questionnaire and its subscales
MIQ-3 total score | 2 years
  MIQ-3 total score was got after calculate the all values.

SECONDARY OUTCOMES:
MIQ-3 subscale score | 2 years
  MIQ-3 subscore was got after calculate the all values for each subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)